CLINICAL TRIAL: NCT04702152
Title: The Role of Context in Sleep-related Memory Reactivation in Humans: the Effects of Direct Context Reactivation During Sleep on Memory
Brief Title: The Effects of Direct Context Reactivation During Sleep on Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Eitan Schechtman-Drayman, Postdoctoral Fellow at the Cognitive Neuroscience Lab, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00213443-A
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Sleep; Consolidation
MeSH Terms: interventions — Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): This is a within-subject study with a single group of participants
  Interventions: Behavioral: Targeted memory reactivation (sounds)

INTERVENTIONS:
Behavioral: Targeted memory reactivation (sounds) — I will unobtrusively and repeatedly present learning-related sounds during sleep using speakers. This method was shown to improve memory in various tasks. The sounds will be presented several seconds apart and the volume will be so adjusted as not to disturb the participant's sleep. The sounds will be presented during non-rapid eye movement sleep (sleep stage 2 and slow wave sleep). The sounds presented will be non-congruently related to the scenes in the previous learning task. This manipulation is within-subject - all participants will get it, but different specific sounds will be presented for each individual participant.

SUMMARY:
The context in which memories are encoded is a major factor influencing how memories are organized. Individual memories are bound to the context (e.g., the location, time and state of mind in which they are encoded) and this context is later reinstated to recall the details related to the memory. Although the role of context has been explored with regard to memory encoding and retrieval, its role during sleep-related memory consolidation has not been explored. Memories are thought to be reactivated during sleep, subsequently benefitting from the process. This study will use encephalography (EEG) in humans to consider several competing hypotheses regarding context's role in sleep reactivation, thereby enhancing the current understanding of how reactivation of memory over sleep relates to models of context and memory. Participants will learn to associate pictures of scenes to different sounds and to smaller images of items and animals, and then learn the spatial locations of these smaller images on a grid. Crucially, for half of these scenes, the sounds themselves will then also be linked directly to some of images during training. The associated sounds will then be unobtrusively presented during sleep, in a manner that has been shown to improve associated memories. The subsequent memory benefits will reveal whether (1) all images associated with the cued scene will benefit from cuing, demonstrating a context-reactivation effect; (2) only the images directly associated with presented sound will benefit from the cuing, demonstrating a item-reactivation effect; or (3) some composite of these two models. Regardless of which hypothesis is correct, the results will expand our current understanding regarding the role context plays in sleep consolidation.

DETAILED DESCRIPTION:
Each participant will be run in a single afternoon, which includes a 90-minute nap opportunity. Before the nap, participants will go through training and test sessions - and after it they will partake of final memory tests. Neural activity will be continuously monitored and recorded throughout the task using electrophysiological equipment.

This is a within-subjects study. The main manipulation is the unobtrusive presentation of sounds during sleep, a technique called targeted memory reactivation (TMR). All participants will hear these sounds, but the specific sounds each one will hear will be different. The results will then be compared within participant, not between different groups or individuals. Appropriate statistical methods for such analyses include paired t-test and repeated measures analysis of variance. The choice of which sounds will be presented to each participant will be made based on their performance in the pre-sleep test. This will be done in an attempt to balance pre-sleep scores between presented and unpresented stimuli to remove statistical noise. Both the participant and the experimenter will be blind to which sounds will be presented, and the selection will be automatically made by the computer. This technique has been extensively used and has no known risks.

There are two main reasons that using a within-subject design reduces the required sample size. First, the lack of a between-subject independent variable intuitively requires less participants. Second, the level of statistical noise due to individual differences is reduced (i.e., because each participant is compared with their own scores). Previous TMR studies, which have found significant cuing effects, commonly used 20-25 participants. I plan to include at least 30 participants in this study, after omitting participants who could not complete the task and those who were not sufficiently cued during sleep. Having 30 participants will allow the use of more powerful statistical methods (in accordance with the common rule of thumb derived from the central limit theorem, which states that means based on sample sizes of more than 30 participants can be assumed to follow a normal distribution). I expect the context-related TMR effect (see summary) to be smaller in magnitude relative to the common effect size observed in spatial learning TMR studies (Hedge's g = 0.39 based on a recent meta-analysis). This is why I included a higher sample size. It is important to note that even if this benefit will be of a smaller magnitude, as I expect, it will still be indicative of the underlying neurocognitive process and therefore extremely valuable for our mechanistic understanding of the role of context in sleep. Aiming at a sample size of at least 30 participants and assuming an omission rate of 80%, I therefore plan to have 38 participants altogether.

Here is a brief summary of the procedure:

Stimuli: 16 images of spatial scenes (e.g., a beach) will each be arbitrarily associated with a sound and with four smaller images of objects or animals. Half of the scenes will be randomly designated to the context-reactivation (CR) condition and half to the item-reactivation (IR) condition (see below). The 64 images will each have a unique 2D position on a circular grid presented on the screen.

Training: Participants will first learn to associate each scene with the paired sound up to criterion. Next, they will learn to associate the scene with its four images up to criterion. The last part of training will include two type of learning blocks that will be interspersed. During the spatial-training blocks, in each trial participants will have to place a single image in its correct location. They will then receive feedback to improve. The scene associated with the image will be presented while they learn, but crucially the sound will never be presented for the CR condition scenes. For the IR scenes, the sound will be presented while learning two of the items, but never for the other two.

An alternative design might have divorced the cued items in the CR condition from the scenes altogether; the items could have been associated with novel sounds (i.e., that were not connected to the scene) and not presented along with their scene. However, using such a design would have introduced a confounding factor. The novel sound may have still been associated, to an unknown degree, not only to the item but also to the context to which it belongs. The degree to which this novel sound would be associated with the context would therefore remain uncontrolled and may vary between participants and scenes. Sounds used for item in the IR condition are always additionally associated with the scene. By always having the sounds be associated both with context and - in the IR condition - additionally to items, I substantially reduce any interpretation issues.

During the Sound-scenes blocks, which do not include a spatial component or the smaller images at all, the scenes will be presented with the sounds only for the CR condition scenes (i.e., to balance the number of sound presentations between conditions). These blocks will repeat in an interleaved manner until each participant will reach the pre-set learning criterion on the spatial-task.

Pre-sleep test: After training, participants will be tested on their spatial-memory for all items without exposure to sounds or scenes.

Sleep: During NREM (non-rapid eye movement) sleep, the sounds associated with half of the CR condition scenes and half of the IR condition scenes will be presented unobtrusively. The choice of which sounds to present will be made in a manner that will balance pre-sleep results and therefore enhance the contrast between sleep-related effects for cued and non-cued images.

Post-sleep test: At least 10 minutes after the end of the nap, participants will undergo a test identical to the pre-sleep one. Immediately after, they will be tested on the scene-item and scene-sound associations using both a free-recall and a recognition test. Participants will then be thanked, debriefed, paid and dismissed.

ELIGIBILITY:
Inclusion Criteria:

---

Exclusion Criteria:

Participants with a history of neurological disorders or of sleep disorders will be excluded.

Participants who do not believe they would be able to fall asleep in the lab will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in error rates between pre- and post-sleep for the different conditions | Approximately 15 minutes before sleep onset and approximately 15 minutes after sleep offset within the same experimental session
  The correct location of an image is compared with the position in which the participant has placed it. Measured in pixels on a computer screen.
Modulation of EEG spectral power following sound/odor presentation | During sleep within the experimental session, assessed up to 1.5 hours
  Power modulations within the sigma (12-16 Hz), theta (4-8 Hz) and delta (0.5-4 Hz) ranges immediately following sound onset. Measured across different EEG channels.

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuroscience Lab - Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No